CLINICAL TRIAL: NCT06251089
Title: Randomized, Double-blind, Multicenter Pilot Clinical Trial to Evaluate the Use of a Mouthwash With Cetylpyridinium Chloride (CPC) in the Prevention and Reduction of Symptoms of Viral Upper Respiratory Tract Infections (vURTI)
Brief Title: Effect of Cetylpyridinium Chloride (CPC) Rinse in Viral Upper Respiratory Tract Infections (vURTI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentaid SL (Industry)
Collaborators: Methodex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MTH_DEN0123
Record Dates: First submitted 2024-01-08; First posted 2024-02-09 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-02

CONDITIONS: Viral Pharyngitis
Keywords: CPC; viral upper-respiratory infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.07% CPC mouthwash (Experimental): Brush your teeth twice a day with fluoride toothpaste, after meals. Then rinse for 1 minute with 15 ml of the test mouthwash for 1 minute. If feasible on the part of the volunteer, they will be asked to do 30 seconds of gargling and 30 seconds of mouthwash.
  If the volunteers are unable to rinse, the health professionals who care for them will be asked to perform the application of the product using sterile gauze soaked with the product, passing it through the oral mucous membranes and tongue, twice a day
  Interventions: Drug: CPC mouthwash
- comparator (Placebo Comparator): Brush your teeth twice a day with fluoride toothpaste, after meals. Then rinse for 1 minute with 15 ml of the control product for 1 minute. If feasible on the part of the volunteer, they will be asked to do 30 seconds of gargling and 30 seconds of mouthwash.
  If the volunteers are unable to rinse, the health professionals who care for them will be asked to perform the application of the product using sterile gauze soaked with the product, passing it through the oral mucous membranes and tongue, twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CPC mouthwash — 0.07% CPC mouthwash
  Arms: 0.07% CPC mouthwash
Drug: Placebo — placebo of the CPC mouthwash
  Arms: comparator

SUMMARY:
This is a randomized, controlled clinical trial with two parallel groups in which 150 volunteers (75 per group) will receive either VITIS CPC Protect® mouthwash (Mouthwash with cetylpyridinium chloride (CPC) as an anti-plaque antiseptic at a concentration of 0.07%) or mouthwash without cetylpyridinium chloride, as control group Subjects included in the study will be followed for 90 days. Symptoms associated with vURTIs (viral upper respiratory tract infections) should be recorded, when they appear, to determine the existence of viral infections of the upper respiratory tract.

Symptoms and adverse effects will be recorded when the episode occurs. The assignment as VURIs will be made by the investigator once the diaries have been completed, or during the symptoms if possible.

DETAILED DESCRIPTION:
This is a randomized, controlled clinical trial with two parallel groups in which 150 volunteers (75 per group) will be included. Allocation ratio (1:1). The trial will be offered to subjects who live in a nursing home and who can perform mouthwashes themselves or to whom healthcare professionals can apply the product.

Subjects included in the study will be followed for 90 days. Symptoms associated with vURTI should be recorded, when they appear, to determine the existence of viral infections of the upper respiratory tract. If such an infection exists (when three of the following symptoms are present: fever over 37º, non-productive cough, sore throat, runny nose, nasal congestion or malaise) the degree of severity will be determined and recorded.

Symptoms and adverse effects will be recorded when the episode occurs. The assignment as vURTI will be made by the investigator once the diaries have been completed, or during the symptoms if possible. Follow-up visits will be conducted fortnightly

ELIGIBILITY:
Inclusion Criteria:

* Subjects admitted to nursing home
* Subjects who have had a washing period of 2 months since the last use with mouthwashes.
* > age 65
* Subjects who are able to do mouthwashes or receive oral hygiene by caregivers
* Delivery of the Participant Information Sheet (HIP) and signing of the Informed Consent (IC) to subjects or legal guardians of the subjects who agree to participate.

Exclusion Criteria:

* Subjects who are suffering from an upper or lower airway infection at the time of recruitment
* Subjects who are physically or psychologically unable to perform mouthwashes or receive oral hygiene with gauze or cotton soaked in antiseptic
* Subjects who have used oral antiseptics continuously in the past month
* Use of oral hygiene measures outside the study conditions
* Subjects who frequent residences, but are not admitted (e.g. day centre) Subjects or legal guardians of subjects who do not provide their IC to participate Subjects who have a registered allergy to the product or to the excipients of the product.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
occurrence of vURTI episodes | 3 months
  the occurrence or non-occurrence of vURTI episodes. VURI is considered when three of the following symptoms are present: Fever over 37º; Non-productive cough; Sore throat; Rhinorrhoea; Nasal congestion; Discomfort

SECONDARY OUTCOMES:
description of vURTI | 3 months
  number of vURTI
description of vURTI | 3 months
  frequency of mild, moderate or severe vURTI
oral health | 3 months
  presence of gingival inflammation,
oral health | 3 months
  presence of mucosal lesions
oral health | 3 months
  presence of plaque

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Blanc, Study Chair — Dentaid SL
Locations (1):
- EAP Baix Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No